CLINICAL TRIAL: NCT02071147
Title: Randomised Trial of Four to Six Week Follow Ups vs no Medical Follow up After Uncomplicated Cataract Extraction
Brief Title: RCT of Follow up Following Cataract Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 14/02/050
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Cataract
Keywords: Follow-up; No follow-up; removal; Randomised Controlled Trial; 6 Weeks
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard clinical intervention (Other): Patients reviewed at 6 weeks (+/- 1 week) as is our normal practice and recalled for a further evaluation if deemed appropriate. Patients will be instructed to visit their optometrist once their eye has fully recovered from the operation for provision of glasses.
  Interventions: Other: Quality of Life questionnaire; Other: Patient satisfaction Questionnaire
- No Clinical Follow up (Other): No routine follow-up appointment is made. Patients will be instructed to visit their optometrist between 6-8 weeks post-operative for review of the patient's glasses.
  Interventions: Other: No Clinical Follow up; Other: Quality of Life questionnaire; Other: Patient satisfaction Questionnaire

INTERVENTIONS:
Other: No Clinical Follow up
  Arms: No Clinical Follow up
Other: Quality of Life questionnaire
  Other Names: VQOL
Other: Patient satisfaction Questionnaire — Conducted at Research clinic.

SUMMARY:
Purpose:

To examine the safety of omitting the routine postoperative eye clinic review following phacoemulsification cataract surgery.

Background:

Approximately 300000 cataract extractions are performed annually in the NHS in England, requiring a similar number of post-operative visits, the majority of which result in no change in management. A conservative estimate of 70% of visits being unnecessary suggests a potential saving to the NHS of approximately £10M annually.

What's involved:

The study involves some questionnaires during the duration of the study. These include questionnaires relating to the quality of life of the patient (conducted before the operation, and at the 3 month research clinic) and a patient satisfaction questionnaire. There is also a research clinic 3 months following the operation.

What are the risks/benefits:

There are no real personal benefits to patients on the trial. The trial aims to provide very important information regarding the safety of discharging patients immediately after surgery. However the trial could potentially save many thousands of unnecessary hospital visits each year.

DETAILED DESCRIPTION:
Method:

The method presented is based on the method employed successfully by one of the applicants in an earlier stuy of the first day postoperative review following cataract surgery which has been peer-reviewed and published in the scientific literature. An earlier draft has been presented to a patient panel and has the benefit of external review by a potential steering group.

Patients undergoing routine elective phacoemulsification cataract surgery will be randomly assigned to either a routine review at 4-6 weeks post-operatively (routine care) or to be discharged from the cataract service immediately post-operatively. All patients will be advised to see their own optometrist at 4-6 weeks for new spectacles if appropriate and will then be reviewed in a research clinic at 3 months post operatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults Aged >= 40 years
* Scheduled for day-case cataract surgery
* Able to give informed consent

Exclusion Criteria:

* Unable to provide written informed consent
* Unable to visit their optometrist post operatively
* Patients with ocular comorbidity that may be affected by cataract surgery or who require monitoring within three months of their operation (including significant diabetic retinopathy, wet age-related macular degeneration (AMD) on treatment, severe/end-stage glaucoma, previous retinal detachment or vitrectomy)
* Patients undergoing another simultaneous ophthalmic procedure
* Patients who suffer from an intra-operative complication requiring early postoperative evaluation (identified at surgery).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Corrected distance visual acuity (VA) | 3 Months
Vision-related quality of life impairment measures are the VCM1 and Catquest questionnaires | 3 Months

SECONDARY OUTCOMES:
Post operative complication rate between the two groups | 3 Months
Post operative patient satisfaction between the two groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Frost, MBchB, MRCP, FRCOphth, PHD, Principal Investigator — Torbay and South Devon NHS Foundation Trust
Locations (1):
- Torbay District General Hospital, Torquay, Devon, United Kingdom